CLINICAL TRIAL: NCT06327633
Title: A Pilot, Prospective, Randomized, Open Label, Parallel, 4-month Study to Explore and Evaluate the Therapeutic Effects of Olfactory Training on the Cognitive Function, Olfactory Function, and Odor-induced Brain Activation in T2DM Patients With Mild Cognitive Impairment.
Brief Title: Effects of Olfactory Training on the Brain Function in T2DM Patients With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZ2024
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes Mellitus; Mild Cognitive Impairment
Keywords: Functional MRI; Cognition; Olfactory training
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction | interventions — Olfactory Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olfactory Training Group (Experimental): The subjects repeatedly sniffed pleasant scents of rose, lemon, clove, eucalyptus, coffee and cinnamon twice a day, 6-min per time, with focus, until the completion of the study. Meanwhile, all patients will also continue on their existing dose and regimen of glucose- lowering schemes throughout the study. Twice weekly phone calls will be performed to evaluate the blood glucose situation, assess the safety of intervention and confirm the compliance of participants.
  Interventions: Other: Olfactory Training
- Control Group (No Intervention): The subjects will maintain the original diet and lifestyle, and also continue on their existing dose and regimen of glucose- lowering schemes throughout the study. Phone calls will be made to evaluate the blood glucose situation.

INTERVENTIONS:
Other: Olfactory Training — The subjects repeatedly sniffed pleasant scents of rose, lemon, clove, eucalyptus, coffee and cinnamon twice a day, 6-min per time, with focus, until the completion of the study.
  Arms: Olfactory Training Group

SUMMARY:
This is a prospective, randomized, open label, parallel, 4-month study to explore and evaluate the therapeutic effects of olfactory training on the cognitive function, olfactory function, and odor-induced brain activation in T2DM patients with mild cognitive impairment (MCI).

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes mellitus;
* Aged: 40 -75 years ;
* Cognitive function assessment suggests mild cognitive impairment;
* A stable glucose-lowering regimen for more than 2 months;
* ≥6 years of education;
* Right-handed.

Exclusion Criteria:

* Cognitive function assessment suggests normal cognition or dementia;
* Other dementia related neurological diseases or depression, Mental dysplasia, mania, schizophrenia, etc in the past 2 years; Central nervous system diseases, including brain trauma, intracranial hemorrhage, acute cerebral infarction, etc;
* Severe sinusitis, nasal cavity and sinus polyps, skull base or nasopharyngeal tumors and other space occupying lesions;
* Congenital diseases and traumatic history of nose, maxillofacial and skull base affecting olfaction.
* With symptoms of upper respiratory tract infection, including nasal congestion, runny nose, fever, etc. on the day of MR examination;
* Diabetic Acute and chronic complications, including diabetic ketoacidosis, diabetic ketoacidosis; a hyperglycemic hyperosmolar state or severe hypoglycemic coma, etc.
* Severe impairment of heart, liver, kidney and other organs;
* Contraindications of MRI examination, such as implantation of metal prosthesis in vivo, claustrophobia, etc;
* Pregnant and lactating women;
* Receive other test drugs currently or within 3 months before participating in the project;
* Known or suspected allergic history to essential oil;
* Taking cognitive-related drugs.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Change of cognitive function (evaluated by MoCA score) | from baseline to 4-month follow-up
  Whether MoCA scores in the two groups of Type 2 diabetes mellitus patients with MCI after intervention were different from those before treatment and the difference of changes between the two groups. The MoCA scale evaluates overall cognitive function, with a total score of 30. Generally, subjects scoring ≥26 points are considered as normal cognition, while between 19-25 points as mild cognitive impairment. An extra point is added If the subject has less than 12 years of education.

SECONDARY OUTCOMES:
Change of olfactory brain activation by fMRI | from baseline to 4-month follow-up
  Whether the activation degree of olfactory task fMRI brain area in the two groups after intervention was different from that before treatment and the difference of changes between the two groups. All patients underwent odor-induced task fMRI on a 3.0T MR scanner with 222 volumes for task fMRI and 230 volumes for resting-state fMRI. The odor-induced task consisted of "fresh air" "rest" and "scent". Odor-induced brain activation was assessed by a general linear model using Statistical Parametric Mapping 12 (SPM12) software. Following extraction of the three separate conditions "fresh air," "scent," and "rest" from the whole sequence, contrasts were made for each participant between "fresh air &gt; rest" and "scent &gt; rest." Odor-induced fMRI data were analyzed in the mask of the olfactory network, including the regions of bilateral parahippocampus, amygdala, piriform cortex, insula, orbitofrontal cortex, hippocampus, and entorhinal cortices.
Change of Olfactory function | from baseline to 4-month follow-up
  Whether the scores of olfactory threshold, identification and memory of the two groups after intervention were higher than those before treatment and the difference of changes between the two groups. Olfactory testing was performed using Olfactory Function Assessment by Computerized Testing (OLFACT) (Osmic Enterprises, Inc.). Based on the University of Pennsylvania Smell Identification Test (UPSIT), OLFACT tests were computerized, standardized, and self-administered. Higher scores indicated better ability to detect odors. Threshold testing was performed by a series of binary dilutions of n- butanol solution in light mineral oil, and scores ranged from 1 to 14. Identification and memory tests included two tasks: task A with 10 different odors, and task B with 20 odors (with 10 same odors in the task A). Each participant was asked to identify each odor from four pictures in tasks A and B and to indicate whether each was old or new in task B. There was a 10-min break in-between.
Change of metabolism | from baseline to 4-month follow-up
  The changes of glycosylated hemoglobin among the two groups before and after intervention. The level of glycosylated hemoglobin <7% means better glucose metabolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhang Z, Zhang B, Wang X, Zhang X, Yang QX, Qing Z, Lu J, Bi Y, Zhu D. Altered Odor-Induced Brain Activity as an Early Manifestation of Cognitive Decline in Patients With Type 2 Diabetes. Diabetes. 2018 May;67(5):994-1006. doi: 10.2337/db17-1274. Epub 2018 Mar 2. PMID 29500313
- [Result] Zhang Z, Zhang B, Wang X, Zhang X, Yang QX, Qing Z, Zhang W, Zhu D, Bi Y. Olfactory Dysfunction Mediates Adiposity in Cognitive Impairment of Type 2 Diabetes: Insights From Clinical and Functional Neuroimaging Studies. Diabetes Care. 2019 Jul;42(7):1274-1283. doi: 10.2337/dc18-2584. Epub 2019 May 21. PMID 31221697